CLINICAL TRIAL: NCT05679063
Title: Therapeutic Exercise and Education in Neurophysiology of Pain in the Quality of Life of Women With Endometriosis: Clinical Trial
Brief Title: Therapeutic Exercise and Education in Neurophysiology of Pain in the Quality of Life of Women With Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Responsible Party: Principal Investigator, Rebeca Abril Coello, Principal investigator, University of Valladolid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EndometriosisCdV2022
Record Dates: First submitted 2022-12-28; First posted 2023-01-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Physical Therapy Modalities; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Trough a randomization program, participants will be assigned to the treatment group or the control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants will not know in which treatment group they are, and the investigator in charge of carrying out the evaluation will not know to which group the subjects he evaluates belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic Exercise and Pain Neurophysiology Education (Experimental): Therapeutic exercise is the systematic and planned execution of posture movements and physical activities to correct or prevent alterations, improve or enhance physical functioning, and prevent risk factors for solid and optimized overall health status.
  Pain Neurophysiology Education:
  Education in pain neurophysiology consists in describing to the patient the neurobiology and neurophysiology of his nervous system pain to improve the processing of it and decrease the threatening meaning of pain.
  Interventions: Other: Physiotherapy
- Sham Comparator (Sham Comparator): Talks about healthy habits
  Interventions: Other: Sham, Control

INTERVENTIONS:
Other: Physiotherapy — A program of therapeutic exercise and education in the neurophysiology of pain will be applied to the participants of the experimental group
  Arms: Therapeutic Exercise and Pain Neurophysiology Education
Other: Sham, Control — Talks about healthy habits
  Arms: Sham Comparator

SUMMARY:
The objective of this study will be to evaluate treatment using ET exercise and pain education in women with endometriosis to achieve improvement in quality of life.

DETAILED DESCRIPTION:
A study will be carried out whose objective is to improve the quality of life in women with endometriosis through a program of therapeutic exercise and education in the neurophysiology of pain. Also as secondary variables will be observed: menstrual symptoms, sexual function, and abdominal wall thickness measured with ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age between 18 and 45 years.
* Women with a medical diagnosis of endometriosis.
* Women with visual analog scale (EVA) between 4 and 10 (moderate-severe pain) during the last 3 months in the suprapubic area, abdomen or perineum both continuously and intermittently.

Exclusion Criteria:

* Women who must have surgery during the study.
* Women who have undergone abdominal or pelvic surgery or who have given birth (vaginal or cesarean) in the last 6 months.
* Women who are pregnant or planning a pregnancy.
* Women with uncorrected pacemakers or coagulopathies, severe comorbid disorder, cancer (in the last 5 years or at present), severe mental disorders, or neuropathies affecting the nerves of the pelvis or lower extremities.
* Physiotherapy treatments or treatments related to pathology or study areas 15 days prior to the beginning of the study.
* Variations in medication in the 3 months prior to the start of the stud

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Woman
Enrollment: 40 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2024-10-12 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in quality of life perception assessed using EUROQuOL 5D - 5L | Baseline, Up to 1 month, Up to 3 months.
  The scale will be administered by one of the researchers, This scale covers five dimensions, each of which is assigned a score from 1 to 5, and with these scores, a code is obtained that indicates the person's quality of life. High values indicate poor quality of life.

SECONDARY OUTCOMES:
Abdominal wall muscle thickness | Baseline, Up to 1 month, Up to 3 months
  The muscle thickness of the abdominal wall with ultrasound according to a defined protocol.
Sexual Function assessed usinf Female Sexual Function Index (IFSF) | Baseline, Up to 1 month, Up to 3 months
  The scale will be administered by one of the researchers. This questionnaire consists of 19 questions and is grouped into six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain; each question has 5 or 6 options, assigning them a score ranging from 0 to 5. The score for each domain is multiplied by a factor and the result final is the arithmetic sum of the domains. A higher score better sexuality
Symptoms associated with menstruation assessed using CVM-22 (quality of life related to menstruation) | Baseline, up to 1 month, up to 3 months
  The scale will be administered by one of the researchers. Minimin value = 0. Maximum value = 66. A high result indicates a good quality of life-related to menstruation

CONTACTS AND LOCATIONS:
Overall Officials: SANDRA JIMENEZ, Doctor, Study Director — University of Valladolid
Locations (1):
- SBFisioterapia, Soria, Soria, Spain